CLINICAL TRIAL: NCT05872360
Title: A Randomized, Double-blind Controlled Trial to Investigate Effects of Amway Bundle Combination of Products on Osteoarthritis & Sarcopenia
Brief Title: To Investigate Effects of Amway Bundle Combination of Products on Osteoarthritis & Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amway (China) R&D Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-SM-09-AY-001
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis; Sarcopenia
Keywords: Amway; Nutrilite Lifestyle; EMS (Electric Muscle Stimulation)
MeSH Terms: conditions — Osteoarthritis; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bundle Group 1 with Nutrilite Lifestyle (Active Comparator): Amway All-plant protein booster: 450g/bottle, containing the following active ingredients and with the guideline of Nutrilite Lifestyle:
  * All-plant protein
  * Peptide
  * HA (hyaluronicacid)
  * Calcium
  * Magnesium
  * Glucosamine
  Facility: EMS (electric muscle stimulation)
  Nutrition Guideline: Nutrilite Lifestyle
  Interventions: Dietary Supplement: Bundle Group 1 with Nutrilite Lifestyle
- Bundle Group 2 without Nutrilite Lifestyle (Active Comparator): Amway All-plant protein booster: 450g/bottle, containing the following active ingredients:
  * All-plant protein
  * Peptide
  * HA (hyaluronicacid)
  * Calcium
  * Magnesium
  * Glucosamine
  Facility: EMS (electric muscle stimulation)
  Interventions: Dietary Supplement: Bundle Group 2 without Nutrilite Lifestyle
- Control Group 1 (Placebo Comparator): Placebo for all-plant protein booster: 450g/bottle, containing the following ingredients: Maltodextrin
  Interventions: Dietary Supplement: Control Group 1
- Control Group 2 with Nutrilite Lifestyle (Placebo Comparator): Placebo for all-plant protein booster: 450g/bottle, containing the following ingredients: Maltodextrin
  Nutrition Guideline: Nutrilite Lifestyle
  Interventions: Dietary Supplement: Control Group 2 with Nutrilite Lifestyle

INTERVENTIONS:
Dietary Supplement: Bundle Group 1 with Nutrilite Lifestyle — All-plant protein booster: 2 spoons (15g), twice per day. Calcium & Magnesium：3 tablets one time per day. Glucosamine: 2 tablets two times per day. 20 minutes training with EMS (Electric Muscle Stimulation) per day. Practice according to Nutrilite Lifestyle Guideline per day.
  Arms: Bundle Group 1 with Nutrilite Lifestyle
Dietary Supplement: Bundle Group 2 without Nutrilite Lifestyle — All-plant protein booster: 2 spoons (15g), twice per day. Calcium & Magnesium：3 tablets one time per day. Glucosamine: 2 tablets two times per day. 20 minutes training with EMS (Electric Muscle Stimulation) per day.
  Arms: Bundle Group 2 without Nutrilite Lifestyle
Dietary Supplement: Control Group 1 — Placebo: 2 spoons (15g), twice per day. Placebo for Calcium & Magnesium：3 tablets one time per day. Placebo for Glucosamine: 2 tablets two times per day.
  Arms: Control Group 1
Dietary Supplement: Control Group 2 with Nutrilite Lifestyle — Placebo: 2 spoons (15g), twice per day. Placebo for Calcium & Magnesium：3 tablets one time per day. Placebo for Glucosamine: 2 tablets two times per day. Practice according to Nutrilite Lifestyle Guideline per day.
  Arms: Control Group 2 with Nutrilite Lifestyle

SUMMARY:
The goal of this interventional study is to evaluate the effects of bundle combination of Amway All-plant protein booster with Nutrilite Lifestyle guideline and/or EMS (Electric Muscle Stimulation) device on Osteoarthritis & Sarcopenia in the middle-aged and elderly (50-70 years old) people.

240 eligible participants will be randomly assigned to 4 equal size study groups (ideally 52 for each group will complete the study) in the two study centers in Shanghai, three site visits will be made during the 6 months of study after screening test. All clinical data will be measured /captured on paper CRF(Case Report Form) and then recorded into CTMS(Clinical Trial Data Management System) for analysis and reporting. It's essential that participants should practice with the assigned guideline and device besides taking the products per day.

Researchers will compare the four groups to see if there is significant improvement of Amway study products with bundle combination of Nutrilite Lifestyle guideline and/or EMS on Osteoarthritis & Sarcopenia in the participants.

ELIGIBILITY:
Inclusion Criteria:

* Chinese males or females, age between 50-70;
* SPPB scale 4 - 9, but walking 400 meters within 15 minutes;
* Reporting <20 min/week in the past month performing regular physical activity and <125 min/week of moderate physical activity;
* Willing to comply with all research requirements and procedures;
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate.

Exclusion Criteria:

* Have used any medication for OA & SA at least one month before this study.
* Subject having done plastic surgery for OA & SA.
* Be involved in any aspect of test administration, i.e., evaluating or overseeing activities related to product.
* Have participated in any clinical study involving the test sites within the previous 6 months, or is subject participating in any clinical study concurrently.
* Have a history of any type of metabolic syndrome, including but not limited to any type of diabetes, obesity and heart disease.
* Have a history of any disease or the presence of health condition on the study sites that the Investigator feels would interfere with the study.
* Be taking antihistamines (> 3x/week) or anti-inflammatory (> 8x/week) on a regular basis, or has the subject taken systemic or topical steroidal medications within 4 weeks of study enrolment.
* Have any of the following conditions or factors that the investigator believes may affect the study objectives caused by medication by protein, glucosamine, calcium and magnesium or supplements to improve capability of the sports.
* Have any allergy caused by all-plant protein and sea-food.
* The regular exercises more than 125 minutes per week.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change of Short Physical Performance Battery (SPPB) score from baseline | baseline day 0, day 180
  Change of Short Physical Performance Battery (SPPB) score [0,12] from baseline to day 180

SECONDARY OUTCOMES:
Change of WOMAC Questionnaire Scores from baseline | baseline day 0, day 90, day 180
  Change of WOMAC Questionnaire Scores from baseline to day 90 and day 180
Change of Visual Analogue Scale/Score (VAS) from baseline | baseline day 0, day 90, day 180
  Change of Visual Analogue Scale/Score (VAS), with range from 0 to 10 (the smaller the score, the better visual result), from baseline to day 90 and day 180
Change of Chalder Fatigue Scale (CFS) from baseline | baseline day 0, day 90, day 180
  Change of Chalder Fatigue Scale (CFS), FS-14, with range from 0 to 14 (the bigger the score, the more fatigue a person feels), from baseline to day 90 and day 180
Improvement of Fat and Muscle Portions measured by Inbody S10 from baseline | baseline day 0, day 90, day 180
  Improvement of Fat and Muscle Portions measured by Inbody S10 from baseline to day 90 and day 180
Change of Hand & Grip Strength measured by Jamar Smart Hand Dynamometer from baseline | baseline day 0, day 90, day 180
  Change of Hand & Grip Strength measured by Jamar Smart Hand Dynamometer from baseline to day 90 and day 180
Change of bone density measured by DXA Bone Densitometer from baseline | baseline day 0, day 90, day 180
  Change of bone density measured by DXA Bone Densitometer from baseline to day 90 and day 180

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Principal Investigator — SPRIM Medical
Locations (2):
- China (2):
  - Raison Healthcare Lab, Shanghai, Shanghai Municipality
  - Raison Healthcare R&D Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basat S, Sivritepe R, Ortaboz D, Sevim E, Atay S, Baygul A. The Relationship Between Osteoarthritis and Sarcopenia in Geriatric Diabetic Patients. Sisli Etfal Hastan Tip Bul. 2021 Dec 29;55(4):516-523. doi: 10.14744/SEMB.2021.42890. eCollection 2021. PMID 35317381
- [Background] Zhong J, Xie W, Wang X, Dong X, Mo Y, Liu D, Yao X, Liu B, Deng W, Su Y, Li Y, Wang X. The Prevalence of Sarcopenia among Hunan Province Community-Dwelling Adults Aged 60 Years and Older and Its Relationship with Lifestyle: Diagnostic Criteria from the Asian Working Group for Sarcopenia 2019 Update. Medicina (Kaunas). 2022 Oct 30;58(11):1562. doi: 10.3390/medicina58111562. PMID 36363519
- [Background] Pickering ME, Chapurlat R. Where Two Common Conditions of Aging Meet: Osteoarthritis and Sarcopenia. Calcif Tissue Int. 2020 Sep;107(3):203-211. doi: 10.1007/s00223-020-00703-5. Epub 2020 May 18. PMID 32424600
- [Background] De Ceuninck F, Fradin A, Pastoureau P. Bearing arms against osteoarthritis and sarcopenia: when cartilage and skeletal muscle find common interest in talking together. Drug Discov Today. 2014 Mar;19(3):305-11. doi: 10.1016/j.drudis.2013.08.004. Epub 2013 Aug 20. PMID 23973339
- [Background] Matada MS, Holi MS, Raman R, Jayaramu Suvarna ST. Visualization of Cartilage from Knee Joint Magnetic Resonance Images and Quantitative Assessment to Study the Effect of Age, Gender and Body Mass Index (BMI) in Progressive Osteoarthritis (OA). Curr Med Imaging Rev. 2019;15(6):565-572. doi: 10.2174/1573405614666181018123251. PMID 32008564
- [Background] Smith D, Knapp PK, Wright DC, Hollick DR. Dual Energy X-Ray Absorptiometry (DXA) Extended Femur Scans to Support Opportunistic Screening for Incomplete Atypical Femoral Fractures: A Short Term in-vivo Precision Study. J Clin Densitom. 2023 Apr-Jun;26(2):101352. doi: 10.1016/j.jocd.2022.12.005. Epub 2022 Dec 8. PMID 36740545
- [Background] Lee SY, Choo PL, Pang BWJ, Lau LK, Jabbar KA, Seah WT, Chen KK, Ng TP, Wee SL. SPPB reference values and performance in assessing sarcopenia in community-dwelling Singaporeans - Yishun study. BMC Geriatr. 2021 Mar 30;21(1):213. doi: 10.1186/s12877-021-02147-4. PMID 33781211
- [Background] Marcos-Pardo PJ, Gonzalez-Galvez N, Carbonell-Baeza A, Jimenez-Pavon D, Vaquero-Cristobal R. GDLAM and SPPB batteries for screening sarcopenia in community-dwelling Spanish older adults: Healthy-age network study. Exp Gerontol. 2023 Feb;172:112044. doi: 10.1016/j.exger.2022.112044. Epub 2022 Dec 9. PMID 36509296
- [Background] Petrella RJ, DiSilvestro MD, Hildebrand C. Effects of hyaluronate sodium on pain and physical functioning in osteoarthritis of the knee: a randomized, double-blind, placebo-controlled clinical trial. Arch Intern Med. 2002 Feb 11;162(3):292-8. doi: 10.1001/archinte.162.3.292. PMID 11822921
- [Background] Doshi R, Ostrovsky D. Glucosamine may be Effective in Treating Pain due to Knee Osteoarthritis. Explore (NY). 2019 Jul-Aug;15(4):317-319. doi: 10.1016/j.explore.2019.04.007. Epub 2019 May 4. No abstract available. PMID 31229448
- [Background] Train A, Moe S, Allan GM. Are glucosamine and chondroitin natural remedies for osteoarthritis? Can Fam Physician. 2021 Feb;67(2):111. doi: 10.46747/cfp.6702111. No abstract available. PMID 33608362
- [Background] Angelides S, Manolios N. Correspondence on 'Glucosamine and O-GlcNAcylation: a novel immunometabolic therapeutic target for OA and chronic, low-grade systemic inflammation?'. Ann Rheum Dis. 2023 Mar;82(3):e57. doi: 10.1136/annrheumdis-2020-219694. Epub 2021 Jan 27. No abstract available. PMID 33504484
- [Background] Welch C, Majid Z, Greig C, Gladman J, Masud T, Jackson T. Interventions to ameliorate reductions in muscle quantity and function in hospitalised older adults: a systematic review towards acute sarcopenia treatment. Age Ageing. 2021 Feb 26;50(2):394-404. doi: 10.1093/ageing/afaa209. PMID 33098419
- [Background] Wakabayashi H, Sakuma K. Comprehensive approach to sarcopenia treatment. Curr Clin Pharmacol. 2014 May;9(2):171-80. doi: 10.2174/1574884708666131111192845. PMID 24219006